CLINICAL TRIAL: NCT04829578
Title: A Prospective Study of Hypnosis for Chronic Idiopathic Pruritus
Brief Title: Hypnosis for Chronic Idiopathic Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-AOIP-01; 2020-A03263-36 (Other: CHU de Nice)
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Idiopathic Pruritus
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypnosis (Other): hyspnosis treatment
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — Chronic idiopathic pruritus is treated by hypnosis

SUMMARY:
Chronic idiopathic pruritus (CIP) is a frequent and disabling condition, for which there is no specific treatment. It was shown previously that hypnosis can relieve painful sensations. Pain and pruritus share many similarities regarding sensory receptors and pathways, suggesting that hypnosis might help relief CIP.

DETAILED DESCRIPTION:
Chronic idiopathic pruritus (CIP) is a frequent and disabling condition, with significative impact on quality of life. At present, there is no specific treatment for CIP. Topical steroids are frequently used, with partial efficacy, and adverse effects. Hypnosis is a specific state of conscience. It differs from waking state, sleeping state, relaxation, or meditation. In this state, the person is highly responsive to suggestion. In medicine, hypnosis can be used to engage the internal resources of the person against unpleasant feelings. It was shown previously that hypnosis can relieve painful sensations. Pain and pruritus share many similarities regarding sensory receptors and pathways, suggesting that hypnosis might help relief CIP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 18 years at screening
* Diagnosis of chronic (at least 6 wks.) idiopathic pruritus
* Pruritus Numeric Rating Scale > = 4

Exclusion Criteria:

* Pruritus caused by a dermatological or a systemic conditions
* Suicidal crisis, moderate, or severe
* Psychosis (schizophrenia, persistent delusional disorder)
* Bipolar disorder, not stabilized or decompensating
* Personality disorder, decompensated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pruritus Numeric Rating Scale | Day 84
  Assessment of the intensity of pruritis in Pruritus Numeric Rating Scal; the minimum and maximum values 0 to 10

SECONDARY OUTCOMES:
Change From Baseline in Pruritus Verbal Rating Scale | Day 84
  Assessment of Pruritus by pruritus Verbal Rating Scale; the minimum and maximum values 0 to 4
Change From Baseline in Sleeping Scale | Day 84
  assessment in sleeping scale ; the minimum and maximum values 0 to 10
Change From Baseline in DLQI scale | Day 84
  assessment in DLQI scale; result between 0 to 30
Change From Baseline in HAD scale | Day 84
  assessment in HAD scale; result between 0 to 42
Change From Baseline in usage of topical steroids | Day 84
  assessment in usage of topical steroids
Evaluation of tolerance of hypnosis | Day 84
  assessment of tolerance of hypnosis with report of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: BAHADORAN PHILIPPE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No